CLINICAL TRIAL: NCT04871776
Title: Use of Construal Level Theory to Inform Messaging to Increase Vaccination Against COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nancy Haff, MD, MPH, Associate Epidemiologist, Division of Pharmacoepidemiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021P001308; P30AG064199 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Covid19; Vaccine Refusal
MeSH Terms: conditions — COVID-19; Vaccination Refusal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Why" messaging (Experimental): In this arm, patients will be sent an electronic patient portal message a few days in advance of their office visit. Messages will focus on reasons to get the COVID booster vaccine, including protecting self and loved ones or the idea of herd immunity.
  Interventions: Behavioral: Messaging informed by construal level theory
- "How" messaging (Experimental): In this arm, patients will be sent an electronic patient portal message a few days in advance of their office visit. "How" messages will focus on the details of obtaining a vaccination at MGB, what to expect, and how to prepare for the visit.
  Interventions: Behavioral: Messaging informed by construal level theory
- Usual Care (Active Comparator): In this arm, patients will not receive any additional message about their upcoming visit, beyond what they already receive by the health system.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Messaging informed by construal level theory — Messages are informed by construal level theory, which suggests that emphasizing "why" elicits more abstract thinking, or high-level construals, and can induce an emotional mindset, which could challenge an individual's sense of identity, autonomy, or political preferences. Conversely, emphasizing "how" is more cognitive and evokes concrete thinking, or low-level construals, and encourages a planning or implementation mindset, which may be better for encouraging vaccine uptake.
  Arms: "How" messaging; "Why" messaging
Behavioral: Usual Care — Usual messaging sent by Mass General Brigham
  Arms: Usual Care

SUMMARY:
This study aims to increase uptake of the COVID booster vaccine through messaging informed by Construal Level Theory. Patients in the Mass General Brigham (MGB) health system aged 18 and older who are eligible for the COVID booster vaccine, but who have not yet received a dose at the time of an upcoming primary care clinic visit, will be randomized to one of three messaging arms: 1) "why" messaging, 2) "how" messaging, or 3) standard of care ("usual care"). Messages will be sent via the electronic patient portal a few days in advance of their office visit. The primary outcome will be the rate of booster vaccination at the targeted visit. The secondary outcome will be the rate of receipt of a COVID booster vaccine within 6 weeks of the targeted visit. Subgroup analyses to assess for any association of patient characteristics with intervention responsiveness will be exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the Mass General Brigham system
* Aged 18 and older
* Are eligible for the COVID booster vaccine but have not received a dose at time of upcoming primary care clinic visit

Exclusion Criteria:

* Documented allergy to a COVID vaccine or its components
* Home address outside of Massachusetts
* Did not receive full set of primary COVID-19 vaccination series

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3671 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haff N, Choudhry NK, Bhatkhande G, Keller PA, Robertson T, Oran R, Horn D, Crum KL, Oduol T, Hanken K, Lauffenburger JC. "How" Versus "Why" Messaging to Increase Uptake of Booster Vaccination Against COVID-19: Results of a Pragmatic Randomized Trial. J Gen Intern Med. 2024 Mar;39(4):611-618. doi: 10.1007/s11606-023-08492-x. Epub 2023 Nov 6. PMID 37932539

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The three patient deaths reported here occurred after randomization but before the study intervention could be administered, and so are excluded from primary analyses. In addition, 3 patients were excluded from the primary analysis for not meeting eligibility criteria. Thus the primary analysis consisted of 3665 patients.
Period: Overall Study
Arm/Group | "Why" Messaging | "How" Messaging | Usual Care
Started | 1200 | 1252 | 1219
Completed | 1199 | 1249 | 1217
Not Completed | 1 | 3 | 2
Not completed — Death after randomization but before intervention could have been administered | 0 | 2 | 1
Not completed — Did not meet eligibility criteria | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Six patients were excluded after randomization. The three patients died after randomization but before the study intervention could be administered and three patients were excluded from the primary analysis for not meeting eligibility criteria. Thus the primary analysis consisted of 3665 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | "Why" Messaging | "How" Messaging | Usual Care | Total
Number analyzed (Participants) | 1199 | 1249 | 1217 | 3665
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.23 (17.46) | 53.80 (17.36) | 53.40 (16.96) | 53.5 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 697 | 733 | 736 | 2166
  Male | 502 | 516 | 481 | 1499
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 324 | 322 | 329 | 975
  Not Hispanic or Latino | 769 | 830 | 768 | 2367
  Unknown or Not Reported | 106 | 97 | 120 | 323
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 49 | 48 | 51 | 148
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 74 | 91 | 99 | 264
  White | 724 | 766 | 718 | 2208
  More than one race | 15 | 17 | 17 | 49
  Unknown or Not Reported | 336 | 325 | 332 | 993
Baseline vaccinations, N(%) [Number; unit: participants] — Population: Pneumonia vaccines and zoster vaccines were analyzed only among the populations who would be eligible for those vaccines based on age. Ever received pneumonia vaccine was analyzed among the population age >65 (N = 973). Ever received a zoster vaccine was analyzed among the population age >50) (N = 2101).
  participants
    Flu shot in the past year | 542 | 582 | 537 | 1661
    Ever received pneumonia vaccine (if age >65): number analyzed (Participants) | 324 | 334 | 315 | 973
    Ever received pneumonia vaccine (if age >65) | 287 | 306 | 285 | 878
    Ever received a zoster vaccine *if age >50): number analyzed (Participants) | 682 | 726 | 693 | 2101
    Ever received a zoster vaccine *if age >50) | 329 | 374 | 322 | 1025
    Tetanus vaccine in last 10 years | 962 | 997 | 985 | 2944

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received a Booster Vaccination Through the Targeted Visit
Description: Number of participants who received one dose of a COVID booster vaccine between randomization through the date of the scheduled visit, determined through electronic health records.
Time Frame: 2-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | "Why" Messaging | "How" Messaging | Usual Care
Number analyzed (Participants) | 1199 | 1249 | 1217
Participants | 164 | 146 | 166
Statistical Analysis 1: Comparison: "How" Messaging vs Usual Care; We used generalized estimating equations with a logit link function and binary-distributed errors, adjusting for clinic-day clustering and including clinic as an adjustment variable for all models. This analysis is otherwise unadjusted; Test type: Superiority; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.67 to 1.14] — How vs Usual Care
Statistical Analysis 2: Comparison: "Why" Messaging vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.81 to 1.28]
Statistical Analysis 3: Comparison: "Why" Messaging vs "How" Messaging; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.96 to 1.51]

2. Secondary Outcome: Number of Participants Who Received a Booster Vaccination Within 6 Weeks of the Targeted Visit
Description: Number of participants who received one dose of a COVID booster vaccine between randomization through 6 weeks after the targeted visit, determined through electronic health records.
Time Frame: 6 weeks after the target visit
Measure: Count of Participants; unit: Participants
Arm/Group | "Why" Messaging | "How" Messaging | Usual Care
Number analyzed (Participants) | 1199 | 1249 | 1217
Participants | 264 | 231 | 265
Statistical Analysis 1: Comparison: "How" Messaging vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.67 to 1.01]
Statistical Analysis 2: Comparison: "Why" Messaging vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.87 to 1.23]
Statistical Analysis 3: Comparison: "Why" Messaging vs "How" Messaging; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.06 to 1.49]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between randomization and 6-week follow up for each study participant.
Description: Note that deaths are reported for the randomized sample of 3671. Three deaths occurred after randomization but before intervention could be delivered. These participants were excluded from the primary analytic sample, as indicated in the patient flow section, but the deaths are included here. Two deaths occurred during the 6-week follow up period after primary outcome assessment was complete, also included here. Adverse event data is otherwise presented for the analytic sample of 3665.
Arm/Group | "Why" Messaging | "How" Messaging | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/1200 | 2/1252 | 1/1219
Serious Adverse Events (participants affected / at risk) | 0/1199 | 0/1249 | 0/1217
Other Adverse Events (participants affected / at risk) | 0/1199 | 0/1249 | 0/1217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT04871776/Prot_SAP_000.pdf